CLINICAL TRIAL: NCT02777606
Title: The Efficacy of Si-Ni-Tang (a Chinese Herbal Formula) for Severe Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Lai Fang, Attending Doctor, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014A020212280
Record Dates: First submitted 2016-05-14; First posted 2016-05-19 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Severe Sepsis
Keywords: Severe Sepsis; Sini Decoction; Immune Function; Mortality
MeSH Terms: conditions — Sepsis | interventions — sini tang

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Si-Ni-Tang (a Chinese Herbal Formula) (Experimental): Treatment for severe sepsis adheres to the International guidelines for management of sepsis and septic shock 2012 and the Surviving Sepsis Campaign updated bundles in response to new evidence in 2015. Besides, 150ml of Si-Ni-Tang will be given by p.o. or a nasogastric tube once per day for 3 days in the treatment group.
  Interventions: Drug: Si-Ni-Tang
- Control (No Intervention): Treatment for severe sepsis adheres to the International guidelines for management of sepsis and septic shock 2012 and the Surviving Sepsis Campaign updated bundles in response to new evidence in 2015.

INTERVENTIONS:
Drug: Si-Ni-Tang — Treatment adheres to the International guidelines for management of severe sepsis and septic shock( 2012) and the Surviving Sepsis Campaign updated bundles in response to new evidence in 2015 for both the treatment group and the control group. In addition, 150ml of Si-Ni-Tang will be given by p.o. or by a nasogastric tube once a day for 3 days in the treatment group.
  Other Names: Sini decoction
  Arms: Si-Ni-Tang (a Chinese Herbal Formula)

SUMMARY:
The purpose of this study is to evaluate the efficacy of Si-Ni-Tang (a Chinese Herbal Formula documented in Shang Han Lun) in treating severe sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Severe sepsis (according to American college of chest Physicians/ Society of Critical Care Medicine (ACCP/SCCM) criteria)
* Informed consent provided by patients or legally authorized representative
* Yin syndrome in syndrome differentiation (according to principles of traditional Chinese medicine (TCM) syndrome differentiation)

Exclusion Criteria:

* Pregnant or nursing female
* Subject receiving immunosuppressive or immunoenhancement therapy in the past 3 months
* Patients with known or suspicious autoimmune diseases
* Patients not expected to survive 28 days due to end-stage disease or other uncorrectable medical condition
* Fasting subjects
* Known or suspicious allergy to any ingredient of Si-Ni-Tang
* Patients not expected to survive 5 days for various reasons

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
28-day all-cause mortality rates | 28 days after enrollment
  28 days all-cause mortality rates after enrollment

SECONDARY OUTCOMES:
Human leukocyte antigen DR (HLA-DR) expression on cluster of differentiation (CD) 14 T lymphocytes | day 0 and 3after enrollment
  HLA-DR expression on cluster of differentiation (CD) 14 T lymphocytes measured on day 0 and 3 after enrollment
CD 4+/ CD 8+ ratio | day 0 and 3after enrollment
  CD 4+/ CD 8+ ratio measured on day 0 and 3 after enrollment
procalcitonin (PCT) | day 0 and 3 after enrollment
  PCT measured on day 0 and 3 after enrollment
Sequential Organ Failure Assessment (SOFA) score | day 0 and 3 after enrollment
  SOFA score measured on day 0 and 3 after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Fang Lai, Master, Principal Investigator — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zeng R, Zheng Y, Fan R, Zhou G, Zhang Y, Mai S, Xie D, Weng Y, Du J, Han Y, Lai F. Si-ni-tang (a Chinese herbal formula) for improving immunofunction in sepsis: study protocol for a pilot randomized controlled trial. Trials. 2019 Aug 28;20(1):537. doi: 10.1186/s13063-019-3646-3. PMID 31462310